CLINICAL TRIAL: NCT03318081
Title: The Application of Cognitive Rehabilitation Therapy for Amphetamine-type Stimulants Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MZhao-008
Record Dates: First submitted 2017-10-15; First posted 2017-10-23 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Amphetamine Addiction
Keywords: Amphetamine-type stimulants; prefrontal-striatal circuits; cognitive rehabilitation therapy
MeSH Terms: conditions — Amphetamine-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cognitive function rehabilitation group (Active Comparator): The main content of cognitive function rehabilitation esecutive function,including working memory,sustained attention, response inhibition function and cognitive flexibility, 45 minutes a day over 6 weeks period.
  Interventions: Behavioral: cognitive function rehabilitation and bias modification
- cognitive bias modification group (Active Comparator): The main content of cognitive bias modification groups were changing ATS related attention bias, 45 minutes a day over 6 weeks period.
  Interventions: Behavioral: cognitive function rehabilitation and bias modification
- control group (No Intervention): Participants only accept the regular scheduled in the compulsory isolated detoxification center

INTERVENTIONS:
Behavioral: cognitive function rehabilitation and bias modification — cognitive rehabilitation focus on the deficits executive funcitin and elevated cognitive bias
  Arms: cognitive bias modification group; cognitive function rehabilitation group

SUMMARY:
The computerized cognitive rehabilitation therapy will be used to treat amphetamine-type stimulant (ATS) addiction.

DETAILED DESCRIPTION:
The deficits in executive functions related to prefrontal-striatal circuits play a vital role in ATS addiction and relapse, and proposed computerized cognitive rehabilitation therapy as the novel interventions. Focused on evaluating and training executive functions including working memory, inhibitory control, cognitive flexibility, and congitive bias concerning prefrontal-striatal circuits, neuropsychological tests, electroencephalography tests, magnetic resonance spectroscopy (MRS) and functional MRI will be used to evaluate the therapeutic effect of ATS addiction treatment as well as investigate the mechanisms. The study will be very helpful to develop novel interventions in clinical practice and decrease ATS-related harm for both the patients and their families.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed MA dependence in accordance with the fourth edition of the American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) (Association, 2000);
2. more than 9 years of education;
3. aged of 18-60 years old;
4. normal vision, audition and no color blindness;
5. receive no detoxification medications during treatment and
6. right handedness.

Exclusion Criteria:

1. current medical diseases that required hospitalization or regular monitoring;
2. serious physical or neurological illness that required pharmacological treatment affecting cognitive function;
3. history of major psychiatric disorder such as bipolar disorder, schizophrenia, depression and disorders of high comorbidity with substance abuse/dependence;
4. neurological diseases such as stroke, seizure, migraine, head trauma
5. substance dependence other than nicotine, within the past 5 years;
6. intelligence quotient (IQ) <70.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Craving for ATS assessed by Visual Analog Scales (VAS) at 1 month , 3 month and 6 months | Baseline, 1 month, 3 month and 6 months
  evaluate all participants' craving for ATS by Visual Analog Scales (VAS): The scores of the VAS were 0-10 points. 10 points reflect the highest level of individual's craving, and 0 point reflect no craving in patient.

SECONDARY OUTCOMES:
Cognitive function assessed by CogState Battery (CSB) | Baseline, 1 month, 3 month and 6 months
  evaluate all participants' cognitive function by the computerized CogState Battery (CSB) Chinese version: The five tasks listed below were examined. International shopping list task (ISLT, verbal learning and memory), the score is defined as the total number of correct responses. Continuous paired association learning task (CPAL) taps spatial working memory. Groton maze learning task (GML) taps problem solving/error monitoring. The scores of CPAL and GML tasks are the total number of errors. Social emotional cognition task (SEC, social cognition) asks the subjects to pick out the different facial expressions. Two back task (TWOB, working memory) requires subjects to decide whether a card is identical to the one shown just before. The scores of TWOB and SEC tasks are the proportion of correct responses, denoting the accuracy of performance. The higher values represent a better outcome in ISL, SEC and TWOB. The higher values represent a worse outcome in GML and CPAL.
Changing of response inhibition ablility assessed by Balloon Analogue Risk Task (BART) | Baseline, 1 month, 3 month and 6 months
  evaluate all participants' response inhibition function by Balloon Analogue Risk Task (BART): Several indices were computed to represent the behavioral performance, including the ratio of all pumps to numbers of win trials, the ratio of pumps to numbers in win trials, and the number of win trials. The higher values represent a worse outcome.
Number of participants who relapse | 1 month, 3 month and 6 months
  Follow up with patients after discharge, evaluate number of participants who relapse. The higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Min, PhD, MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Compulsory Isolation Detoxification Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu Y, Jiang H, Su H, Zhong N, Li R, Li X, Chen T, Tan H, Du J, Xu D, Yan H, Xu D, Zhao M. A Newly Designed Mobile-Based Computerized Cognitive Addiction Therapy App for the Improvement of Cognition Impairments and Risk Decision Making in Methamphetamine Use Disorder: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Jun 20;6(6):e10292. doi: 10.2196/10292. PMID 29925497